CLINICAL TRIAL: NCT06627803
Title: Multi-Method Investigation of Social Facilitation of Alcohol Effects and Alcohol Misuse in Young Adults
Brief Title: Social Facilitation of Alcohol Effects and Alcohol Misuse in Young Adults
Acronym: PALS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Matthew Kirkpatrick, Associate Professor, University of Southern California
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: UP-24-00590; 1R01AA031240-01A1 (NIH)
Record Dates: First submitted 2024-10-02; First posted 2024-10-04 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Alcohol Consumption; Alcohol Abuse/Dependence
MeSH Terms: conditions — Alcohol Drinking; Alcoholism | interventions — Ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Laboratory alcohol administration with longitudinal follow-ups (Experimental): All participants will be in this single arm, which consists on behavioral testing of alcohol administration in the lab, followed by longitudinal follow-ups using Ecological Momentary Assessment and surveys.
  Interventions: Drug: Alcohol (Oral)

INTERVENTIONS:
Drug: Alcohol (Oral) — Participants will drink a beverage that will have alcohol or no alcohol. The amount of alcohol consumed will be similar to consuming around 3-4 drinks, with breath alcohol concentration peaking at or around the legal limit for driving (0.08%).

SUMMARY:
The purpose of this study is to understand social contexts and alcohol use. We hope to learn how being around peers affects alcohol consumption in young adults. About 200 young adults who drink alcohol frequently will take part in the study. This research is being funded by the National Institute on Alcohol Abuse and Alcoholism (NIAAA).

Participation involves one in-person screening session with a same-sex platonic friend. Then participants will complete four in-person laboratory sessions where they will drink beverages containing alcohol or no alcohol. After completion of the laboratory sessions, participants will complete smartphone surveys for 28 days. Lastly, they will complete follow-up surveys 6 months and 12 months post-study enrollment.

ELIGIBILITY:
Inclusion Criteria:

* 21-28 years of age
* Drink regularly (1+ times/week) with a same-sex platonic friend that also meets eligibility and is willing to participate
* Regular alcohol use (3+ times/week) with at least one binge drinking episode (5+ drinks [male] or 4+ drinks [female] in about 2 hours) in the past month
* BMI of 18-30
* Own a smart device operating on the iOS or Android operating system
* Fluent in English

Exclusion Criteria:

* Pregnancy or breastfeeding or intent to get pregnant in the next 60 days (females)
* medical conditions counter-indicated for alcohol administration
* seeking treatment for alcohol use

Ages: 21 Years to 28 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-02-20 (Actual); Primary Completion 2029-08-31 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
Drug Effect Questionnaire (DEQ) | The DEQ will be assessed 30 minutes before alcohol administration, and again 30, 60, 90, 120, 180, and 240 minutes after alcohol administration during each session.
  The Drug Effects Questionnaire (DEQ), a 5-item visual analog questionnaire (0 to 100 mm; not at all to extremely), will be used to assess the extent to which participants experience the effects of the drug: "feel drug," "feel high," "like drug," "dislike drug," and "want more".
Biphasic Alcohol Effects Scale (BAES) | The BAES will be assessed 30 minutes before alcohol administration, and again 30, 60, 90, 120, 180, and 240 minutes after alcohol administration during each session.
  The Biphasic Alcohol Effects Scale (BAES) is a 14-item survey that instructs individuals to rate the extent to which drinking alcohol has produced related subjective effects (0=not at all to 10=extremely). This questionnaire has two subscales consisting of mean scores related to sedation and stimulation.
Quantity of Alcohol Use during Ecological Momentary Assessment | Quantity of Alcohol Use will be assessed daily for 28 days.
  Quantity of alcohol use will be the number of drinks reported each day during the Ecological Momentary Assessment period. Number of drinks reported will be recoded to create two binary variables alcohol use (alcohol use [1+ drinks], no alcohol [0]) and binge drinking (binge [female: 4+ drinks; male: 5+ drinks], no binge (female: <4 drinks; male<5 drinks]).
Past 30-day Alcohol Use during Follow-Up | Past 30-day alcohol use will be assessed 6 and 12 months after the initial laboratory sessions.
  Past 30-day alcohol use (including number of drinks and binge drinking) will be assessed using the timeline follow-back method.

SECONDARY OUTCOMES:
Positive and Negative Affect Schedule (PANAS) | The PANAS will be assessed 30 minutes before alcohol administration, and again 30, 60, 90, 120, 180, and 240 minutes after alcohol administration during each session.
  The Positive and Negative Affect Schedule (PANAS) is a well-validated brief scale comprised of 20 items meas-uring positive affect (e.g., excited, inspired) and negative affect (e.g., upset, afraid) in the moment. Each item is rated on a five-point Likert Scale, ranging from 1 = Very Slightly or Not at all to 5 = Extremely).
Brief Young Adult Alcohol Consequences Questionnaire (YAACQ) during Ecological Momentary Assessment | The YAACQ will be completed daily for 28 days.
  The validated Brief Young Adult Alcohol Consequences Questionnaire (YAACQ) is a 24-item measure assessing negative alcohol-related consequences. Summary scores are the sum of all items.
Past 30-day Alcohol Consequences during Follow-Up | Past 30-day alcohol consequences will be assessed at 6 and 12 months following the initial laboratory sessions.
  Past 30-day alcohol consequences will be assessed using the validated Brief Young Adult Alcohol Consequences Questionnaire (YAACQ), a 24-item measure assessing negative alcohol-related consequences. Summary scores are the sum of all items.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Per NOT-AA-22-003, this study will submit and share de-identified demographic and primary and secondary outcome data with NIAAA Data Archive (NIAAADA), a data repository housed within the NIMH Data Archive (NDA). Datasets will be findable and identifiable through a persistent study digital object identifier (DOI) generated by NDA.
Supporting Information: Study Protocol
Time Frame: We will submit data on or before the NDA submission due dates (April 1 and October 1 each year of the award starting in 2025) in accordance with the applicable Data Sharing Terms and Conditions of award. We will perform QA/QC checks on data within 4 months after the submission due dates and address any issues identified by the NDA.
  Study data will be available to the research community in perpetuity. Additionally, upon acceptance of a manuscript for publication, we will submit to NIAAADA data used in that publication to allow future analysts to replicate and expand upon the results.
Access Criteria: All study data will be deidentified and thus will be made available as public use data to the research community via NIAAADA. Users of the public use data must register with the NIAAADA data archive and agree to the Terms of Use, which are designed to protect study participants by limiting data use to scientific research and aggregate statistical reporting, prohibiting attempts to identify study participants, and requiring immediate reporting of any disclosure of study participant identity.